CLINICAL TRIAL: NCT04919174
Title: A Randomized Single-blind Clinical Trial of the Efficacy and Safety of Remimazolam in Painless Bronchoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0058
Record Dates: First submitted 2021-05-24; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-04

CONDITIONS: Bronchoscopy; Sedation
Keywords: remimazolam, dexmedetomidine, bronchoscopy, sedation
MeSH Terms: interventions — remimazolam; Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Patients receive dexmedetomidine for sedation
  Interventions: Drug: Dexmedetomidine
- Test group (Experimental): Patients receive remimazolam for sedation
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Sedation with remimazolam
  Other Names: Remifentanil
  Arms: Test group
Drug: Dexmedetomidine — Sedation with dexmedetomidine
  Other Names: Remifentanil
  Arms: Control group

SUMMARY:
Over the past decade, bronchoscopy technology has developed rapidly and has become an important part of the diagnosis and treatment of respiratory diseases. Bronchoscopy are usually carried out under monitored anesthesia care (MAC), which can relieve the anxiety of the patient, make the operation easier, and improve the completion rate of bronchoscopy. At present, bronchoscopy has widely used midazolam, propofol, short-acting opioids, and newer sedatives such as dexmedetomidine, but each drug has its limitations. Dexmedetomidine is widely used in non-intubation general anesthesia and sedation during short outpatient surgery. However, rapid and high-dose infusion of dexmedetomidine leads to dose-dependent hypotension, temporary hypertension, bradycardia, and excessive sedation, causing hemodynamic fluctuations. At the same time, it has slow onset and metabolism. This may be a potential risk for some elderly patients with many underlying diseases and unstable hemodynamics. Remimazolam is an ultra-short-acting benzodiazepine. It has the advantages of short action time, low accumulation, low risk of respiratory depression, and reversibility. We believe that remimazolam can improve the onset time and resuscitation time, to achieve sufficient sedation, improve the success rate of bronchoscopy, while reducing the patient's oxygen saturation drop during the operation, postoperative opioid-related nausea and vomiting, postoperative delirium and other related adverse events. This study is a randomized controlled trial to confirm the above hypothesis.

DETAILED DESCRIPTION:
All patients undergoing bronchoscopy under general anesthesia will be recruited and should complete relevant preoperative examinations. The patient fasted for 6-8 hours before the operation, and an indwelling trocar was placed in the vein. After entering the room, the patient will be monitored with electrocardiogram(ECG), pulse oximetry, non-invasive blood pressure, and underwent oxygen inhalation (5L/min) through a nasal cannula. All patients used 2% lidocaine glue to moisten the nasal cavity for local anesthesia before the operation, the bronchoscope was inserted through the nose. The subjects take a supine position. When the bronchoscope passes through the vocal cords and carina, 5 ml of 2% lidocaine is delivered through the channel to suppress the cough reflex. Then the patients were randomly divided into two groups:

1. one group use dexmedetomidine-remifentanil for anesthesia: the initial dose of dexmedetomidine is 0.1ml/kg, infused for 5 minutes, and then adjusted to 0.1-0.5ml/kg/h; the initial dose of remifentanil is 0.05ml/kg, infused for 5 minutes, and then adjusted to 0.1- 0.5 ml/kg/h.
2. the other group use remimazolam-remifentanil for anesthesia: the initial dose of remimazolam is 0.1ml/kg, infused for 5 minutes, and then adjusted to 0.1-0.5ml/kg/h; the initial dose of remifentanil is 0.05ml/kg, infused for 5 minutes, and then adjusted to 0.1- 0.5 ml/kg/h.

All patients started bronchoscopy when they reached TE sedation (modified observer's assessment of sedation,MOAA/S score 3 points). If the assessment of sedation after administration suggests that the sedation is insufficient, propofol 0.4-0.6 mg/kg is repeatedly administered every 5 minutes, with the maximum dose not exceeding 200 mg to maintain sedation. In the maintenance phase of sedation, appropriate sedation is pre-defined as a MOAA/S score of 4 or less. The drug was continuously infused until the end of the bronchoscopy, and all patients were transferred to the post-anaesthesia care unit (PACU) for further observation.

Data from the DoCare Clinic electronic anesthesia recording system was used in this experiment. Bronchoscopy was performed by the same bronchologist with more than 10 years of experience.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 years old.
2. Need for bronchoscopy (for example, unexplained cough, hemoptysis, localized wheezing and hoarseness, chest X-ray and/or CT scans suggest abnormalities, examination and evaluation of lungs before surgery, chest trauma, lungs Or bronchial infectious disease).
3. ASA classification I-III level.
4. BMI≤30kg/m2.
5. Women of childbearing age have a negative pregnancy test.
6. Before the study, the patients voluntarily signed and dated the informed consent form approved by the institutional review board.

Exclusion Criteria:

1. Patients with known allergies to benzodiazepines, flumazenil, opioids, naloxone or certain drugs.
2. Patients with long-term use of benzodiazepines or opioids.
3. Patients with a history of drug abuse or alcohol abuse in the past two years.
4. Bradycardia (baseline HR <60bpm) or hypotension (baseline SAP<100mmHg).
5. Asthma or chronic obstructive pulmonary disease(COPD) or FEV1<1.0L.
6. SpO2 <90% before bronchoscopy.
7. Patients who received any study drug within 30 days before screening or less than 7 half-lives of the drug.
8. Any patient with cognitive impairment or inability to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Decreased Oxygen Saturation [ Safety] | Within 1 hour after the operation
  Oxygen Saturation<90%, more than 30s
Interruption Rate of Bronchoscopy [effectiveness] | Within 1 hour after the operation
  the occurrence of body movement or coughing makes the operating physician have to suspend the operation for physical restraint or adding drugs

SECONDARY OUTCOMES:
Blood Pressure | Within 1 hour after the operation
  Hemodynamic variable
Heart Rate | Within 1 hour after the operation
  Hemodynamic variable
Hemodynamic variable | Within 1 hour after the operation
  SpO2
Respiratory Rate | Within 1 hour after the operation
  Hemodynamic variable
Anesthesia onset time | Within 1 hour after the operation
  onset time (min)
Remedial drug demand dose of the two groups of patients | Within 1 hour after the operation
  Remedial drug demand dose
Satisfaction Scores of The Operating Physicians | Within 1 hour after the operation
  Satisfaction Scores (0-5,higher scores mean a better outcome.)
Incidence of adverse reactions | Within 1 hour after the operation
Incidence of operation-related complications | Within 1 hour after the operation
Anesthesia resuscitation time | Within 1 hour after the operation
  resuscitation time (min)

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, MD, Study Chair — Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No